CLINICAL TRIAL: NCT05819047
Title: Assessment of Upper Limb Motor Performance Using an Interface With Haptic Feedback
Status: Completed | Type: Observational
Sponsor: Universidad Nacional de Entre Rios (Other)
Responsible Party: Principal Investigator, Rosa María Weisz, Principal Investigator, Universidad Nacional de Entre Rios
Other Study IDs: IS003960
Record Dates: First submitted 2023-04-05; First posted 2023-04-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: Haptic technology; Musculoskeletal pain; Virtual environment
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy: Healthy volunteers
  Interventions: Device: Functional test with a haptic device

INTERVENTIONS:
Device: Functional test with a haptic device — Volunteers will complete two tests based on the Nine Hole Peg Test with a haptic device.

SUMMARY:
The purpose of the study is to test an evaluation environment based on a device that has the ability to provide the user with tactile (haptic) sensations. This environment will be used to investigate how the arm movements of a healthy person are performed, and then - at a later stage - to find out whether it is possible to measure changes during musculoskeletal pain. Electrical signals produced by the brain (called electroencephalogram or EEG) will be recorded by means of electrodes on the surface of the scalp (non-invasive). In addition, the angle of the elbow joint during movement will be measured, with the intention of using objective measures to aid future evidence-based clinical decision making.

It is expected that the developed environment can be used -in the near future-, to evaluate the progression of pathologies associated with muscle pain, or to quantify the effectiveness of rehabilitation therapies.

DETAILED DESCRIPTION:
Experimental setup Volunteers will be received at the Center of Rehabilitation Engineering and Neuromuscular and Sensory Research (CIRINS). They will be informed, in simple terms, of the purpose of the project and the measurements that will be done during the session. The Informed Consent Form will be read to each volunteer and, if they decide to participate, they will be asked to sign a copy that will be filed in the Laboratory together with their contact information, which will be stored confidentially.

At the beginning of the session, the volunteer will be asked to sit comfortably. The EEG electrodes will then be attached using a 16-electrode cap in the standard 10-20 location, together with the exoskeleton in the position determined by the investigator. The position of the camera that will be used to follow the movements of the upper limb will also be adjusted to ensure that the movements will be within the camera's field of view.

Subsequently, the subject will be placed in its initial position: seated, with approximately 45° of shoulder abduction, 10° of shoulder flexion and 90° of elbow flexion.

Once the subject is in the proper position, they will be asked, using the implemented test interface, to perform the virtual nine-hole peg test (NHPT) in Cue Based and Self Paced variants. The volunteer will be asked to complete these tests with both hands, in order to assess whether there are differences in performance associated with the side with which the test is performed, and whether using the system is sensitive enough to detect these changes. The researcher conducting the experiment should record which test was performed with the dominant hand and which was not.

To evaluate whether the results obtained are satisfactory, they will be compared with those reported for healthy individuals.

Evaluation tests Cue-based nine-hole peg test: this test works with time or event dependent cues, dividing the test into several repetitions of the same task. Each trial starts at the same predetermined position, and consists of placing as quickly as possible a random peg in a random hole. This randomness is given in the order of the first nine attempts without repeating the peg. Then, in case of additional attempts, the order of the first nine attempts is repeated. In case of failure to complete an attempt within a certain time or placing the peg in the wrong hole, it is given as failed. The signals presented to the user are visual. The pegs change color from white (inactive) to red, which marks the peg that should move (but without giving the signal to move yet), when the peg changes to green, the movement should begin. Likewise, the hole into which the peg should be inserted is marked with the addition of a translucent light blue object. Inactive holes have no color or object inside. At the end of a repetition, the position of the pegs is reset. The starting point of each repetition of the test is marked with a translucent sphere, which is the position that the robot cursor must take before the next attempt. This object sees its position reflected along with the other elements of the virtual environment when changing hands.

Self-paced nine-hole peg test : this test gives the user the freedom to place the desired peg in the desired hole at the desired speed. This test is the most similar to the original NHPT, and ends when all nine pegs are placed in the nine holes, giving as a result the total duration of the test.

ELIGIBILITY:
Inclusion Criteria:

* No history of neurological disease, chronic pain, or musculoskeletal disorders.
* Willingness and ability to fully understand the content and scope of the experiment and to comply with the instructions.
* Signature of the informed consent document.

Exclusion Criteria:

* Pregnancy.
* History of chronic pain or neuromuscular disorders.
* History of addictive behavior, defined as abuse of alcohol, cannabis, opioids or other drugs.
* History of heat sensitivity disorders.
* Presence of fever, tuberculosis, malignant tumors, infectious processes, acute inflammatory processes.
* Implantation of pacemakers or metallic prostheses.
* Use of analgesics within 24 hours prior to participation in the experiment.
* Lack of cooperation.
* Trauma of the segment to be evaluated in the last 4 weeks.
* Surgical history of the upper quadrant.
* Metabolic diseases.
* Ingestion of pain medication in the last 24 hs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Movement smoothness | Average of 36 trials during a single experimental session with a duration of 30 minutes
  Smoothness of the participant movement calculated through the fourth derivative of the trajectory (jerk).

SECONDARY OUTCOMES:
Log jerk transport | Average of 36 trials during a single experimental session with a duration of 30 minutes
  Smoothness of the peg transport trajectory, from the initial position to the hole.
Log jerk return | Average of 36 trials during a single experimental session with a duration of 30 minutes
  Smoothness of the return trajectory, from the position of the hole where the last peg was inserted to the initial position of the next peg.
SPARC return | Average of 36 trials during a single experimental session with a duration of 30 minutes
  Smoothness of the return trajectory, from the position of the hole where the last peg was inserted to the initial position of the next peg.
Path length ratio transport | Average of 36 trials during a single experimental session with a duration of 30 minutes
  Efficiency of the peg transport trajectory, from the initial position to the hole.
Path length ratio return | Average of 36 trials during a single experimental session with a duration of 30 minutes
  Efficiency of the return trajectory, from the position of the hole where the last peg was inserted to the initial position of the next peg.
Velocity max. return | Average of 36 trials during a single experimental session with a duration of 30 minutes
  Maximum velocity during the return trajectory, from the position of the hole where the last peg was inserted to the initial position of the next peg.
Jerk peg approach | Average of 36 trials during a single experimental session with a duration of 30 minutes
  Precision of the ballistic movement during the approach to the peg (near the end of the return and just before the beginning of transport).

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Weisz, MSc. in Biomed Eng, Principal Investigator — Universidad Nacional de Entre Rios
Locations (1):
- Facultad de Ingeniería, Universidad Nacional de Entre Ríos, Oro Verde, Entre Ríos Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD except video recordings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The study protocol is available since the protocol registration. IPD, SAP and analytic code will be available 6 months after data collection.
Access Criteria: Open access in a public platform.

REFERENCES:
- [Background] Mista CA, Monterde S, Ingles M, Salvat I, Graven-Nielsen T. Reorganized Force Control in Elbow Pain Patients During Isometric Wrist Extension. Clin J Pain. 2018 Aug;34(8):732-738. doi: 10.1097/AJP.0000000000000596. PMID 29505418
- [Background] Hodges PW, Tucker K. Moving differently in pain: a new theory to explain the adaptation to pain. Pain. 2011 Mar;152(3 Suppl):S90-S98. doi: 10.1016/j.pain.2010.10.020. Epub 2010 Nov 18. No abstract available. PMID 21087823
- [Background] Karos K, Meulders A, Gatzounis R, Seelen HAM, Geers RPG, Vlaeyen JWS. Fear of pain changes movement: Motor behaviour following the acquisition of pain-related fear. Eur J Pain. 2017 Sep;21(8):1432-1442. doi: 10.1002/ejp.1044. Epub 2017 Apr 25. PMID 28444803
- [Background] Tsay A, Allen TJ, Proske U, Giummarra MJ. Sensing the body in chronic pain: a review of psychophysical studies implicating altered body representation. Neurosci Biobehav Rev. 2015 May;52:221-32. doi: 10.1016/j.neubiorev.2015.03.004. Epub 2015 Mar 14. PMID 25783221
- [Background] Rigsby B, Reed KB. Accuracy of Dynamic Force Compensation Varies With Direction and Speed. IEEE Trans Haptics. 2019 Oct-Dec;12(4):658-664. doi: 10.1109/TOH.2019.2912375. Epub 2019 Apr 23. PMID 31021805
- [Background] Kanzler CM, Schwarz A, Held JPO, Luft AR, Gassert R, Lambercy O. Technology-aided assessment of functionally relevant sensorimotor impairments in arm and hand of post-stroke individuals. J Neuroeng Rehabil. 2020 Sep 25;17(1):128. doi: 10.1186/s12984-020-00748-5. PMID 32977810
- [Background] Kanzler CM, Rinderknecht MD, Schwarz A, Lamers I, Gagnon C, Held JPO, Feys P, Luft AR, Gassert R, Lambercy O. A data-driven framework for selecting and validating digital health metrics: use-case in neurological sensorimotor impairments. NPJ Digit Med. 2020 May 29;3:80. doi: 10.1038/s41746-020-0286-7. eCollection 2020. PMID 32529042
- [Background] Schwarz A, Kanzler CM, Lambercy O, Luft AR, Veerbeek JM. Systematic Review on Kinematic Assessments of Upper Limb Movements After Stroke. Stroke. 2019 Mar;50(3):718-727. doi: 10.1161/STROKEAHA.118.023531. PMID 30776997
- [Background] Wright DJ, Holmes PS, Smith D. Using the movement-related cortical potential to study motor skill learning. J Mot Behav. 2011;43(3):193-201. doi: 10.1080/00222895.2011.557751. PMID 21462065
- [Background] Feys P, Lamers I, Francis G, Benedict R, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. The Nine-Hole Peg Test as a manual dexterity performance measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):711-720. doi: 10.1177/1352458517690824. Epub 2017 Feb 16. PMID 28206826
- [Background] Spuler M, Niethammer C. Error-related potentials during continuous feedback: using EEG to detect errors of different type and severity. Front Hum Neurosci. 2015 Mar 26;9:155. doi: 10.3389/fnhum.2015.00155. eCollection 2015. PMID 25859204
- [Background] J. D. Guzmán, E. F. Fonseca, C. F. Rengifo, D. E. Guzmán, J. Londoño and E. Muñoz, "Implementación de la prueba de funcionalidad motriz de miembro superior nine-hole peg test en un entorno virtual 3D", Iberdiscap, 2017
- [Background] Ahmed T, Thopalli K, Rikakis T, Turaga P, Kelliher A, Huang JB, Wolf SL. Automated Movement Assessment in Stroke Rehabilitation. Front Neurol. 2021 Aug 19;12:720650. doi: 10.3389/fneur.2021.720650. eCollection 2021. PMID 34489855
- [Background] Mista CA, Laugero SJ, Adur JF, Andersen OK, Biurrun Manresa JA. A new experimental model of muscle pain in humans based on short-wave diathermy. Eur J Pain. 2019 Oct;23(9):1733-1742. doi: 10.1002/ejp.1449. Epub 2019 Jul 24. PMID 31251430
- [Background] Gatti R, Atum Y, Schiaffino L, Jochumsen M, Biurrun Manresa J. Decoding kinetic features of hand motor preparation from single-trial EEG using convolutional neural networks. Eur J Neurosci. 2021 Jan;53(2):556-570. doi: 10.1111/ejn.14936. Epub 2020 Aug 25. PMID 32781497
- [Background] W. Wei, "Virtual reality enhanced robotic systems for disability rehabilitation," in Virtual and Augmented Reality: Concepts, Methodologies, Tools, and Applications, 2018
- [Background] S. Mahamad, S. M. Taib, and M. N. Ibrahim, "Analyzing speed accuracy trade-off in control movement mechanism with error enforcement," in Applied Mechanics and Materials, 2011.